CLINICAL TRIAL: NCT07122492
Title: Randomized Controlled Trial of FoRtitude: Targeted eHealth Intervention to Reduce Fear of Recurrence Among Breast Cancer Survivors in Community Oncology Settings
Brief Title: A Targeted Electronic Health Approach to Reduce Fear of Recurrence in Breast Cancer Survivors (FoRtitude)
Acronym: FoRtitude
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: EAQ181
Record Dates: First submitted 2025-08-07; First posted 2025-08-14 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer Survivor; Fear of Cancer Recurrence
Keywords: Breast cancer survivor; Fear of recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): Access to the study intervention website with interactive content, including information to read and videos to watch, and an optional text-messaging feature
  Interventions: Behavioral: FoRtitude 2.0
- Attentive Care (Other): Access to the non-interactive study intervention website that lists links to help you access websites that provide information to read and resources for breast cancer survivors.
  Interventions: Behavioral: Attention Control
- Usual Care (No Intervention): Usual care for fear of recurrence.

INTERVENTIONS:
Behavioral: FoRtitude 2.0 — A website and an interactive text-messaging feature
  Arms: Intervention
Behavioral: Attention Control — Access to the non-interactive study intervention website that lists links to help you access websites that provide information to read and resources for breast cancer survivors.
  Arms: Attentive Care

SUMMARY:
The goal of this study is to determine if the intervention or if general information about being a breast cancer survivor can help Breast Cancer Survivors reduce their fear of recurrence. The main question it aims to answer are:

Can the FoRtitude intervention lower the fear of recurrence for Breast Cancer Survivors?

Participants will:

Answer questions about their fear of recurrence. Be randomized to 1 of the 3 following options: (1) a weblink to access an eHealth intervention which includes a website and an optional interactive text-messaging feature, (2) a weblink to a non-interactive website that will include links to external websites with general information that may be helpful for Breast Cancer Survivors, or (3) you will need to talk with your oncology team about your concerns about recurrence or seek psychosocial care in the community.

Be asked to fill out questionnaires 5 times for up to 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Participant must be ≥ 18 years of age.
* Participant must have had histologically confirmed Stage 0-III breast cancer at time of diagnosis.
* Participant must have completed primary treatment 1-10 years prior to Step 0 registration.

NOTE: Current hormonal therapy is allowed. NOTE: Primary treatment can include chemotherapy and/or surgery and/or radiation therapy.

- Participant must be receiving their care (cancer treatment or survivorship care) from an oncology provider affiliated with the NCORP site and are expected to continue care at the site for the next 18 months.

NOTE: This eligibility criteria is intended to ensure access to healthcare utilization data. Oncology provider can include an Advance Practice Provider, Advance Nurse Practitioner, oncologist, primary care provider, or nurse or physician responsible for survivorship care.

* Participant must have no evidence of active cancer of any type at the time of Step 0 registration (per the assessment of the physician), excluding local basal cell or squamous cell carcinoma.
* Participant must be fluent in written and spoken English.
* Participant must have an ECOG Performance Status of 0-2.
* Participant must have the ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) are not eligible.
* Participant must complete the FCRI 9-item severity scale and report a score of 13 or higher.
* Participant must have access to the internet (via smartphone, tablet, or computer).

NOTE: The restriction to those with internet access is based on the primary intention of the study which involves internet-based delivery intervention content delivered via the internet.

* Participant must have completed the Baseline Assessment within 60 days of Step 0 registration.
* Randomization to Step 1 must occur within 60 days of Step 0 registration.

Exclusion Criteria:

* Participant must not have any psychiatric or cognitive conditions that may affect the participant's ability to accurately provide self-report data, per clinical discretion.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 800 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2028-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
Fear of Cancer Recurrence Inventory (FCRI) | From 1 month post-intervention to 3 months post-intervention
  Fear of Cancer Recurrence Inventory (FCRI) modified total score 143 (without coping or reassurance subscale items) measured during the study period. A graphical exploration of the data will be performed by examining the distribution of FCRI score at each follow up timepoint, as well as the changes in FCRI between the baseline and follow up visits. 1-month post-intervention completion (3 months post-randomization) will be defined as the primary comparison. For the primary analysis we will compare the FCRI score of the FoRtitude arm to each of two control arms at 3 months using Welch's t-test. Two two-group Welch's t-tests will be used to compare the FCRI score of the FoRtitude arm to each of the two control arms at 12 weeks.

SECONDARY OUTCOMES:
Difference in fear of recurrence based on race across all arms | From enrollment to 3 months
  A mixed model, including indicator variables for arm, race, and time, will be used and will include the interactions of race by arm and race by time. The FCRI modified total score of the FoRtitude arm to each of two control arms will be compared at 3 months using a two-group t-test with linear contrasts.
Change in quality of life measures | At all time points, including long term outcomes at 6, 12 and 18 months.
  A per-comparison-wise error rate approach (PCWER) will be used.

CONTACTS AND LOCATIONS:
Overall Officials: Lynne I Wagner, Ph.D., Study Chair — UNC Chapel Hill Gillings School of Global Public Health
Locations (1):
- UNC Chapel Hill School of Medicine Public Health, Chapel Hill, North Carolina, United States